CLINICAL TRIAL: NCT05147792
Title: An Evaluation of the Safety and Effectiveness of the Conformal CLAAS System for Left Atrial Appendage Occlusion
Brief Title: The CONFORM Pivotal Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conformal Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-101
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CLAAS (Experimental): Transcatheter left atrial occluder
  Interventions: Device: CLAAS
- WATCHMAN / Amulet (Active Comparator): Transcatheter left atrial occluder
  Interventions: Device: WATCHMAN left atrial appendage closure device / Amulet left atrial appendage occluder

INTERVENTIONS:
Device: CLAAS — CLAAS
  Arms: CLAAS
Device: WATCHMAN left atrial appendage closure device / Amulet left atrial appendage occluder — WATCHMAN left atrial appendage closure device / Amulet left atrial appendage occluder
  Arms: WATCHMAN / Amulet

SUMMARY:
The CLAAS® device will be evaluated for safety and efficacy by establishing its performance is non-inferior to the commercially available WATCHMAN® and Amulet™ left atrial appendage closure devices in patients with non-valvular atrial fibrillation. Patients who are eligible for the trial will be randomized to receive either the CLAAS device or the WATCHMAN or Amulet™ devices and will be followed for 5 years after device implant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥18 years
2. Documented non-valvular AF (paroxysmal, persistent, or permanent)
3. High risk of stroke or systemic embolism, defined as CHA2DS2-VASc score of ≥ 3
4. Has an appropriate rationale to seek a non-pharmacologic alternative to long-term oral anticoagulation
5. Deemed by the site investigator to be suitable for short term oral anticoagulation therapy but deemed less favorable for long-term oral anticoagulation therapy.
6. Deemed appropriate for LAA closure by the site investigator and a clinician not a part of the procedural team using a shared decision-making process in accordance with standard of care
7. Able to comply with the protocol-specified medication regimen and follow-up evaluations
8. The subject (or legally authorized representative, where allowed) has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate institutional review board (IRB)/Regional Ethics Board (REB)/Ethics Committee (EC).

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to one year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Anatomic conditions that would prevent performance of an LAA occlusion procedure (e.g., atrial septal defect (ASD) requiring closure, high-risk patent foramen ovale (PFO) requiring closure, a highly mobile inter-atrial septal aneurysm precluding a safe TSP, presence of a PFO/ASD closure device, history of surgical ASD repair or history of surgical LAAO closure)
3. Atrial fibrillation that is defined by a single occurrence or that is transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
4. A medical condition (other than atrial fibrillation) that mandates long-term oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or prosthetic mechanical heart valve)
5. History of bleeding diathesis or coagulopathy, or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated
6. Documented active systemic infection
7. Symptomatic carotid artery disease (defined as >50% stenosis with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is <50% stenosis noted at the site of prior treatment
8. Recent (within 30 days of index procedure) or planned (within 60 days post-procedure) cardiac or major non-cardiac interventional or surgical procedure
9. Recent (within 30 days of index procedure) stroke or transient ischemic attack
10. Recent (within 30 days of index procedure) myocardial infarction
11. Vascular access precluding delivery of implant with catheter-based system
12. Severe heart failure (New York Heart Association Class IV)
13. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any prosthetic mechanical valve implant
14. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation)
15. Platelet count <75,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3
16. Known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium) that would preclude any P2Y12 inhibitor therapy, or the patient has contrast sensitivity that cannot be adequately pre-medicated
17. Actively enrolled or plans to enroll in a concurrent clinical study in which the active treatment arm may confound the results of this trial
18. Unable to undergo general anesthesia
19. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 5 years
20. A condition which precludes adequate transesophageal echocardiographic assessment

Echo exclusion criteria:

1. Left atrial appendage anatomy which cannot accommodate a commercially available control device or the CLAAS Implant per manufacturer IFU (e.g., the anatomy and sizing must be appropriate for both the investigational (CLAAS) and a commercially available device in order to be enrolled in the trial)
2. Intracardiac thrombus or dense spontaneous echo contrast consistent with thrombus, as visualized by TEE prior to implant
3. Left ventricular ejection fraction (LVEF) <30%
4. Moderate or large pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology
5. Atrial septal defect that warrants closure
6. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (excursion >15 mm or length > 15 mm) or large shunt (early [within 3 beats] and/or substantial passage of bubbles, e.g., >20)
7. Moderate or severe mitral valve stenosis (mitral valve area <1.5 cm2)
8. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch
9. Evidence of cardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Procedure-related complications, all-cause death, major bleeding | 12 months
  The primary safety endpoint is a composite of 1) major procedure-related complications including a) cardiac perforation, b) pericardial effusion requiring drainage, c) ischemic stroke, d) device embolization, and e) major vascular complications, or 2) major bleeding, or 3) all-cause death
Ischemic stroke and systemic embolism | 18 months
  The primary effectiveness endpoint is a composite of ischemic stroke and systemic embolism through 18 months.

SECONDARY OUTCOMES:
All Cause Mortality | 18 months
  A secondary safety endpoint is all-cause mortality including cardiovascular through 18 months
Myocardial Infarction | 7 days
  A secondary safety endpoint is myocardial infarction evaluated through 7 days post-procedure
Neurologic Events | 45 days
  A secondary safety endpoint is neurologic events including stroke (ischemic and hemorrhagic) and TIA
Closure Success | 12 months
  A secondary performance and efficacy endpoint is closure success at 12 months based upon each of the following criteria: a) demonstration of peri-device leak </=5 mm, and b) demonstration of peri-device leak </=3 mm

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, M.D., Principal Investigator — Lankenau Heart Institute; Shephal Doshi, M.D., Principal Investigator — Pacific Heart Institute
Locations (82):
- United States (70):
  - Grandview Medical Center, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Pima Heart & Vascular, Tucson, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Loma Linda University Health, Loma Linda, California
  - Huntington Hospital, Pasadena, California
  - Pacific Heart Institute, Santa Monica, California
  - Community Memorial Hospital Ventura, Ventura, California
  - Hartford Health Care St. Vincent's Medical Center, Bridgeport, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Ascension St. Vincent's Jacksonville, Jacksonville, Florida
  - Largo Medical Center, Largo, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Baptist Health Care - Pensacola, Pensacola, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - AdventHealth Tampa, Tampa, Florida
  - USF - Tampa General Hospital, Tampa, Florida
  - Piedmont Health Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Inc, Atlanta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Ascension St. Vincent - Carmel, IN, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Terrebone - Cardiovascular Institute of the South, Houma, Louisiana
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Lahey Hospital & Medical Centeer, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford St. John Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Henry Ford Providence Southfield Hospital, Southfield, Michigan
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Cardiac Arrhythmia Research, LLC, Overland, Missouri
  - CHI Health / CommonSpirit Research Institute, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cooper University - Heart House, Haddon Heights, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Albany Medical Center / Capital Cardiology Associates, Albany, New York
  - University of Buffalo / Kaleida Health, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - TriHealth, Cincinnati, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Legacy Emanuel Hospital and Health, Portland, Oregon
  - UPMC Harrisburg, Mechanicsburg, Pennsylvania
  - Lankenau Heart Institute, Wynnewood, Pennsylvania
  - Lifespan Health System, Providence, Rhode Island
  - Prisma Health, Columbia, South Carolina
  - Trident Medical Center, North Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist, Houston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - CHRISTUS Health, Tyler, Texas
  - Senatra Norfolk, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Bellin Health, Green Bay, Wisconsin
- Nemocnice Na Homolce, Prague, Czechia
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHU La Timone, Marseille, Marseille
  - Institut Cardiovasculaire Paris Sud, Massy
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse, Toulouse
- Georgia (4):
  - Chapidze Heart Disease Center, Tbilisi
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - Tbilisi Heart Center, Tbilisi
- Uzbekistan (2):
  - Republican Specialized Center for Surgery named after V. Vakhidov, Chilanzar, Tashkent
  - AKFA Medline, Olmazor, Tashkent

IPD SHARING:
Plan to Share IPD: No